CLINICAL TRIAL: NCT06632366
Title: The Effect Of Awareness-Based Self-Compassage Educatıon Gıven To Women Experıenced Sexual Dysfunctıon In The Postpartum Perıod On The Qualıty Of Sexual Lıfe And Partnershıp
Brief Title: The Effect of Self-Compassion Training on Sexual Life Quality and Marital Adjustment in Women With Sexual Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Fadime BİÇER ŞAHİN, lecturer, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17; Hacer ÜNVER KOCA (Other: ınönü univercity)
Record Dates: First submitted 2024-04-26; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Postpartum Sexual Dysfunction
Keywords: postpartum, midwifery, sexuality
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Intervention Model Description: This research was designed as a randomized controlled experimental type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual Dysfunction in the Postpartum Period (Experimental): In the research, Awareness-Based Self-Compassion Training sessions will be held with the women in the experimental group twice a week for 3 weeks, six times in total.Women in the postpartum period included in the control group will be interviewed twice in total. In the first interview, the "Personal Information Form", "Sexual Life Quality Scale-Female" and "Male Compatibility Scale" will be applied and pre-test data will be obtained. Eight weeks after the pre-test data is obtained, post-test data will be obtained by applying the "Arizona Sexual Experiences Scale-Female", "Sexual Quality of Life Scale-Female" and "Dutch Compatibility Scale".
  Interventions: Other: Sexual Dysfunction in the Postpartum Period
- control (No Intervention): Women in the postpartum period included in the control group will be interviewed twice in total. In the first interview, the "Personal Information Form", "Sexual Life Quality Scale-Female" and "Male Compatibility Scale" will be applied and pre-test data will be obtained. Eight weeks after the pre-test data is obtained, post-test data will be obtained by applying the "Arizona Sexual Experiences Scale-Female", "Sexual Quality of Life Scale-Female" and "Dutch Compatibility Scale".

INTERVENTIONS:
Other: Sexual Dysfunction in the Postpartum Period — The experimental group will receive mindfulness-based self-compassion training. The control group will not receive any intervention.
  Arms: Sexual Dysfunction in the Postpartum Period

SUMMARY:
Sexual function in the postpartum period, the gateway to newness and change, can be affected by problems such as caring for a new baby, breastfeeding, fatigue, anxiety about pain during sexual intercourse, postpartum depression, pelvic floor dysfunction, urinary symptoms and body image. Changes in sexual function are common in the postpartum period. Pregnancy and childbirth is a period in a woman's life that causes hormonal and physical changes and has an impact on the parents' quality of life.

Postpartum sexual function is an important issue for couples, as the first sexual intercourse after childbirth is an important step for couples to establish intimate relationships. Many factors affect postpartum sexual dysfunction, including number of births, breastfeeding, mode of delivery, episiotomy, physical and psychological dysfunction, including fatigue and postpartum depression. Without adequate information and counseling on sexual life by health professionals in the postpartum period, most women may remain silent about their sexual concerns and anxieties, preferring instead to share their problems with friends. More holistic and multidisciplinary approaches are needed to treat female sexual dysfunctions. The use of mindfulness-based therapies has recently become widespread in the treatment of women diagnosed with sexual dysfunction.Thanks to mindfulness practices, it has been observed that women perceive stimuli better and are able to notice clues that they did not notice before. The Compassion Focused Therapy program is one of these practices. It is known to integrate well with existing approaches to therapy and offers some useful ways of reducing sexual problems to provide a coherent rationale for treatment strategies.

DETAILED DESCRIPTION:
The postpartum period is a 6-12-week period that starts with the delivery of the placenta and continues with the disappearance of the physiologic and anatomic changes that occurred during pregnancy . Spousal and family support is very important for a healthy and harmonious passage of this period. With the realization of delivery, the mode of delivery, body image changes, hormonal changes, lactation and breast problems, fatigue, vaginal bleeding, problems related to the baby, sexual reluctance and the relationship between spouses affect the sexual life of women. Although the time to start postpartum sexual intercourse varies from person to person and culture to culture, this period is traditionally 6 weeks. As a result of the studies, it is reported that the time to start postpartum sexual intercourse is between 5-8 weeks. Couples are concerned about starting sexual intercourse when there is bleeding, laceration or episiotomy in the woman in the postpartum period. Physiologic changes that occur during pregnancy and delivery affect sexual intercourse in the postpartum period, and perineal pain and dyspareunia due to episiotomy and laceration are observed in women. However, according to studies, sexual function problems encountered by women in this period include dyspareunia, pelvic floor dysfunction, vaginal dryness, sexual desire / intercourse. satisfaction as a decrease in sexual satisfaction. In a study conducted by Lagaert et al. with 109 women in the postpartum period; women who had spontaneous vaginal delivery and women who had interventional delivery were compared and women who had interventional delivery stated that they experienced more painful sexual intercourse . In the postpartum period, reasons such as episiotomy, perineal pain, vaginal bleeding and discharge, fatigue, pelvic floor dysfunction, feeling less attractive due to physical changes lead to a decrease in sexual desire and consequently to withdrawal from sexuality.

During the first year after birth, new parents face many personal and interpersonal changes, including changes in their sexual relationships. In particular, it has been found that most new parents experience sexual concerns specific to the postpartum period, wondering when to restart sexual intercourse after birth, pain during sexual intercourse, and the impact of body image concerns on sexual activity. Lorenz et al. found that couples generally experienced a decrease in the frequency of sexual activity in the postpartum phase . In a study conducted with 1507 women in the postpartum period, 89% of women were reported to have sexual health problems. In the postpartum 3rd month, the most common complaints were loss of sexual desire, pain during sexual intercourse, and vaginal dryness. Although traditional and complementary treatment practices are utilized in the treatment of sexual dysfunctions, the effectiveness of very few of them has been shown in studies with high level of evidence. Traditional and Complementary Medicine practices used in sexual dysfunctions include natural products (plants, vitamins, minerals and probiotics etc.), mind and body practices such as yoga, mindfulness-based intervention, acupuncture and other methods. The use of mindfulness-based therapies has recently become widespread in the treatment methods of women diagnosed with sexual dysfunction. With these therapies, it has been observed that there is a significant improvement in general sexual function level, arousal and sexual problems. Through mindfulness practices, it has been observed that women perceive stimuli better and are able to recognize clues that they did not notice before. Compassionate mindfulness program is one of these practices. CFT (Compassion Focused Therapy) is known to integrate well with existing approaches to psychosexual therapy and offers some useful ways to reduce sexual problems to provide a coherent rationale for treatment strategies .Self-compassion proceeds in parallel with the individual's self-knowledge, acceptance, positive perspective towards life, social activities, consciousness, character structure open to development and subjectivity. There is an inverse relationship with anxiety disorder, mental depression and the negativities provided by negative situations.

In order to develop compassionate involvement in therapy, the therapist's non-judgmental, warm and encouraging stance when talking about sexual intercourse, as well as detailed information about sexual difficulties, can be a starting point for the client to cope with the difficulties they experience. The therapist can then use a normalizing and non-shaming CFT (Compassion Focused Therapy) formulation to help the client turn towards the difficulties they are experiencing and look at them with understanding. In this sense, the place of midwives who are in constant one-to-one communication with women in the protection and development of sexual health is very important. Determining the sexual needs of women in any period of women's life, eliminating sexual problems, explaining behaviors and attitudes related to sexual life, providing education and guidance are among the roles of midwifery. Midwives have the responsibilities of taking anamnesis, identifying sexual problems and providing education and counseling for these problems in order to maintain and increase the sexual health of pregnant women during pregnancy. It is important for midwives to communicate as a very good listener, to take into account the concerns of the woman, to ask effective questions, to speak by reassuring and stating that privacy will be ensured, to identify the sexual problems of the woman and to provide effective counseling.

ELIGIBILITY:
Inclusion Criteria:

* Erbal communicator and no literacy disability,
* Living with his wife,
* Beginning postpartum sexual intercourse, menstrual cycle has not started
* Between 2-6 months postpartum,
* Having a healthy baby
* Menstrual cycle has not started
* Women diagnosed with sexual dysfunction (total score ≥19) according to the Arizona
* Sexual Experiences Scale will be included in the study.

Exclusion Criteria:

* Having undergone gynecological surgery during the study,
* Have been or are currently diagnosed with a psychiatric illness,
* Having attended any awareness-based training at least 6 months ago

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — postpartum women
Enrollment: 108 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Arizona Sexual Experiences Scale- Female (ASES-F) | ten weeks
  The female form includes questions investigating sexual drive, psychological arousal, physiological arousal (vaginal lubrication), the capacity to reach orgasm and the feeling of satisfaction after orgasm. Each question in the scale is scored from 1 to 6, and the minimum score that can be obtained from the total score is 5 and the maximum is 30. A total score of 19 and above from the scale, a score of 5 or 6 for any item or a score of 4 for three or more items indicates the presence of sexual dysfunction. While low scores represent that the sexual response is effective, comfortable and satisfying, high scores indicate the presence of sexual dysfunction. The total internal consistency coefficient of the scale is 0.89 and the Cronbach alpha reliability coefficient is 0.90.

SECONDARY OUTCOMES:
Sexual Quality of Life Scale- Female (SQOL-F) | ten weeks
  The reliability level of the scale was determined to be high and the reliability coefficient of the scale and the Cronbach alpha value are equal to each other and are 0.83. The scale, which consists of a total of 18 questions, requires answers to problems related to sexual life, including the last 4 weeks. The scale is Likert-type and has a six-point response option. The scoring system of the scale is between 0 and 5 or 1 and 6. The minimum and maximum score that can be obtained from the scale is 18-108. In addition, when the scale is scored between 0 and 5, the score range is 0-90. High scores obtained from the scale indicate that the quality of sexual life is good. The reliability of the scale, which has a reliability coefficient and Cronbach alpha value of 0.83, is high.

OTHER OUTCOMES:
The Revised Marital Adjustment Scale | ten weeks
  The scale was developed to evaluate the relationship quality of married or cohabiting couples in marriage or similar dual relationships. The 7th, 8th, 9th, and 10th items of the scale are reverse scored. The highest score that can be obtained from the scale is 70 points, the obtained score indicates the relationship quality. The Cronbach alpha coefficient of the YÇUÖ with three sub-dimensions is .87, .80, .80, .74 for the total score, satisfaction, consensus, and consensus sub-scales, respectively. The correlation of the scale with the Marital Adjustment Scale used for criterion-dependent validity was calculated as 68 (p<0.01) in the positive direction (Busby et al. 1997).

CONTACTS AND LOCATIONS:
Overall Officials: Hacer Ünver Koca, PhD, Study Director — İnönü University
Locations (1):
- Gaziantep Provincial Directorate of Health, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolsoy N, Sen S, Sezer G, Cakil M. The effect of training on women with postpartum sexual dysfunction: A randomized controlled trial. Niger J Clin Pract. 2023 Jul;26(7):949-956. doi: 10.4103/njcp.njcp_656_22. PMID 37635579
- [Background] De Souza A, Dwyer PL, Charity M, Thomas E, Ferreira CH, Schierlitz L. The effects of mode delivery on postpartum sexual function: a prospective study. BJOG. 2015 Sep;122(10):1410-8. doi: 10.1111/1471-0528.13331. Epub 2015 Mar 6. PMID 25752211
- [Background] Bhat GS, Shastry A. Sexually Induced Orgasm to Improve Postpartum Pelvic Floor Muscle Strength and Sexual Function in Primiparous Women After Vaginal Delivery: A Prospective Randomized Two-Arm Study. J Sex Med. 2022 Nov;19(11):1634-1643. doi: 10.1016/j.jsxm.2022.08.189. Epub 2022 Sep 25. PMID 36167664
- [Background] Kolberg Tennfjord M, Hilde G, Staer-Jensen J, Siafarikas F, Engh ME, Bo K. Effect of postpartum pelvic floor muscle training on vaginal symptoms and sexual dysfunction-secondary analysis of a randomised trial. BJOG. 2016 Mar;123(4):634-42. doi: 10.1111/1471-0528.13823. Epub 2015 Dec 22. PMID 26691895